CLINICAL TRIAL: NCT01705951
Title: Effect of Resistance Training on Tobacco-Related Cardiovascular Disease Risk
Acronym: START
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California (Other)
Responsible Party: Principal Investigator, Christian Roberts, PhD, Research Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 19KT-0028; UL1TR000124 (NIH)
Record Dates: First submitted 2012-10-05; First posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Smoking; Cardiovascular Disease Risk
Keywords: Smoking; Insulin resistance; Metabolic Syndrome; Endothelial Function; Smoking Cessation; Resistance Training; Nicotine Replacement; Exercise; Cardiovascular Disease; Arterial Stiffness; Body Composition
MeSH Terms: conditions — Smoking; Insulin Resistance; Metabolic Syndrome; Smoking Cessation; Motor Activity; Cardiovascular Diseases | interventions — Resistance Training; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Resistance Training/Nicotine Replacement (Experimental)
  Interventions: Other: Resistance Training (RT); Biological: Nicotine Replacement Therapy (NRT)
- Group 2: Resistance Training only (Experimental)
  Interventions: Other: Resistance Training (RT)
- Group 3: Nicotine Replacement Therapy only (Experimental)
  Interventions: Biological: Nicotine Replacement Therapy (NRT)
- Group 4: Control; no RT and no NRT (No Intervention)

INTERVENTIONS:
Other: Resistance Training (RT) — Resistance Training program 3x/week at 60 minutes per session for 12 weeks.
  Arms: Group 1: Resistance Training/Nicotine Replacement; Group 2: Resistance Training only
Biological: Nicotine Replacement Therapy (NRT) — Nicotine patch for 12 weeks (21mg, 14mg, 7mg.) and referral to California Smoker's Helpline for 6 sessions of smoking cessation counseling.
  Other Names: GlaxoSmithKline Nicoderm CQ patch
  Arms: Group 1: Resistance Training/Nicotine Replacement; Group 3: Nicotine Replacement Therapy only

SUMMARY:
This project is prompted by the urgent public health need to identify novel strategies to prevent and treat tobacco-related cardiovascular disease (CVD) and by compelling pilot data that suggests cessation of smoking results in rapid amelioration of endothelial function. The higher prevalence of CVD and metabolic syndrome in smokers have become major health care concerns. Therefore, finding optimal intervention strategies to combat these growing epidemics is imperative. We are investigating the efficacy of resistance training to ameliorate endothelial dysfunction, oxidative stress, inflammation, and insulin resistance in four groups: presence or absence of resistance training with or without cessation treatment + nicotine replacement.

The investigators hypothesize that resistance training will improve cardiovascular function in smokers; however, the responses will be better in those who also stop smoking. In addition, resistance training will decrease smoking, however, the effects of counseling and nicotine replacement alone or counseling and nicotine replacement in conjunction with resistance training will be better than resistance training alone.

DETAILED DESCRIPTION:
The investigators are conducting a 12-week randomized-controlled trial of 100 young adult smokers.

At week 0, participants attend three outpatient visits at baseline. Each participant is randomized to one of four groups: Resistance Training(RT)/Nicotine Replacement Therapy (NRT), RT/No NRT, No RT/NRT, and No RT/No NRT. Those receiving RT work with a certified personal trainer 3 times per week for 12 weeks at 60 minutes each session. Those receiving NRT use the nicotine patch daily for 12 weeks and call the California Smoker's Helpline for smoking cessation counseling. Those in the control group do not receive any intervention and maintain their current lifestyle and habits.

At week 13, participants return for three post-intervention assessments.

At week 26, survey data is collected to assess changes in lifestyle habits.

ELIGIBILITY:
Inclusion Criteria:

* Young Adults (18-35 yrs.)
* Male and female smokers
* Smokers (smoked at least one cigarette a day for 15 or more days in the last month and has smoked 100 cigarettes in life)
* 1-3 years experience consistently exercising/training at ≤2 days/wk of RT and ≤1 day/wk of aerobic exercise
* Capable of providing informed consent
* UCLA students/staff and Non UCLA student/staff
* Participant in good health as determined by baseline visit

Exclusion Criteria:

* Documented CAD
* Has had cardiac surgery
* Currently in weight loss or exercise program in the 6 months prior to participation.
* Use of medications that influence CV function or preclude the ability to train
* Syndromes or prescribed medications that may influence CVD, body composition, or insulin action (e.g. prednisone, Ritalin, Adderall, GH)
* Unable to exercise
* Diagnosed with syndromes or diseases that may influence body composition and CV risk (e.g. Cushing syndrome).
* Known heart arrhythmia and/or abnormalities found in electrocardiogram (ECG) reading that would prevent someone from performing the exercise intervention. If the subject demonstrates abnormal ECG during their pre-intervention visit (or any follow-up visit) the subject's ECG will be reviewed (for approval) by a cardiologist to continue in the study.
* Pregnant
* Use of hormonal contraceptives
* Currently in a smoking cessation program including use of NRT within the month of participation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial function as determined by brachial artery Flow-Mediated Dilation (FMD) | 12 weeks

SECONDARY OUTCOMES:
Smoking cessation percentage | 12 weeks
Arterial stiffness (including PWV and AIx) | 12 weeks
Number of cigarettes smoked | 12 weeks

OTHER OUTCOMES:
Endothelial Progenitor Cells (EPC) count | 12 weeks
  EPC count is measured using a novel flow cytometry protocol.
Insulin sensitivity by Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT) | 12 Weeks
Plasma biomarkers inflammation/oxidative stress (oxidized low density lipoprotein (OxLDL), CRP) | 12 Weeks
Body Composition | 12 Weeks
  Lean mass and fat mass are measured by the Dual Energy X-ray Absorptiometry (DEXA) Scan.
Muscle Strength | 12 Weeks
  Muscle strength is evaluated by a one-Repetition Maximum (1RM) protocol and VO2 peak is assessed by a maximal incremental cardiopulmonary exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Christian K Roberts, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States